CLINICAL TRIAL: NCT00776165
Title: A Phase 3 Randomized Controlled Open Label Comparative Multicentric Trial To Compare The Safety And Efficacy of Indigenous Recombinant Human Granulocyte Colony Stimulating Factor (rhG-CSF) With Neupogen In Patients on Myelosuppressive Therapy for Non Myeloid Malignancies.
Brief Title: Safety and Efficacy Trial of Recombinant Human Granulocyte Colony Stimulating Factor (GCSF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shantha Biotechnics Limited (Industry)
Responsible Party: Dr. Raman Rao, Shantha Biotechnics Limited, Hyderabad, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBL/GCSF/N/2007/0100
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Chemotherapy-Induced Neutropenia
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Recombinant Human Granulocyte Colony Stimulating Factor (rhG-CSF)(Shantha) Dose: 300 mcg/day administered subcutaneous/intravenous/continuous subcutaneous infusion for a minimum of 7 days and for a maximum of 14 days or till Neutrophil count of 10,000/mm3 is reached whichever is earlier
  Interventions: Biological: Recombinant Human GCSF (Shantha Biotechnics Limited)
- 2 (Active Comparator): Neupogen (rhG-CSF) Dose: 300mcg/day administered subcutaneous/intravenous/continuous subcutaneous infusion for a minimum of 7 days and for a maximum of 14 days or till Neutrophil count of 10,000/mm3 is reached whichever is earlier
  Interventions: Biological: Neupogen

INTERVENTIONS:
Biological: Recombinant Human GCSF (Shantha Biotechnics Limited) — Dose: 300 mcg/day administered subcutaneous/intravenous/continuous subcutaneous infusion for a minimum of 7 days and for a maximum of 14 days or till Neutrophil count of 10,000/mm3 is reached whichever is earlier
  Arms: 1
Biological: Neupogen — Dose: 300mcg/day administered subcutaneous/intravenous/continuous subcutaneous infusion for a minimum of 7 days and for a maximum of 14 days or till Neutrophil count of 10,000/mm3 is reached whichever is earlier
  Arms: 2

SUMMARY:
A Phase III Randomized Controlled Open Label Comparative Multicentric Trial To Compare The Safety And Efficacy of Indigenous Recombinant Human Granulocyte Colony Stimulating Factor (rhG-CSF) With Neupogen In Patients on Myelosuppressive Therapy for Non Myeloid Malignancies.

Adult patients (18 years of age or older) diagnosed as having any malignancy (except myeloid malignancy, ECOG status of 0-2 and having a history of experiencing neutropenia (absolute neutrophil count < 1000/mm3) in a previous chemotherapy cycle and have one more cycle of chemotherapy on the same drugs would be recruited into the study.

Treatment will be initiated not earlier than 24 hours after the administration of cytotoxic chemotherapy in both groups.

Group 1: Recombinant Human Granulocyte Colony Stimulating Factor (rhG-CSF)(Shantha)

* Dose: 300 mcg/day administered subcutaneous/intravenous/continuous subcutaneous infusion for a minimum of 7 days and for a maximum of 14 days or till Neutrophil count of 10,000/mm3 is reached whichever is earlier Group 2: Neupogen (rhG-CSF)
* Dose: 300mcg/day administered subcutaneous/intravenous/continuous subcutaneous infusion for a minimum of 7 days and for a maximum of 14 days or till Neutrophil count of 10,000/mm3 is reached whichever is earlier Primary End Point would be to evaluate the percentage of patients developing febrile neutropenia (defined as body temperature ≥ 38.2°C or developing a temperature of > 38°C twice in a 12-hour period and absolute neutrophil count < 0.5 x 109/L on the same day of the fever or the day after)in the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 18 yrs or more
* Patients diagnosed having any malignancy (except myeloid malignancies and myelodysplastic syndromes) receiving standard combination chemotherapy.
* Patients experiencing neutropenia (absolute neutrophil count < 1000/mm3) in a previous chemotherapy cycle and have one more cycle of chemotherapy on the same drugs.
* Patients should have performance status of 0-2 ECOG (European Cooperative Oncology group).

Exclusion Criteria:

* Patients unwilling to give informed consent or unable to follow study procedures
* Patients requiring autologous or allogenic stem cell transplantation.
* Patients having active infection
* Patients who have taken antibiotics or colony stimulation factor within the previous 10 days
* Patients who have clinically significant uncontrolled medical illness except malignancy
* Patients having renal impairment (serum creatinine > 1.5 times the upper normal limit) and abnormal liver function (bilirubin > 5 times the upper limit of normal)
* Pregnant or lactating women
* Patients who have involvement of bone marrow
* Patients receiving simultaneous radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients developing febrile neutropenia (defined as body temperature ≥ 38.2°C or developing a temperature of > 38°C twice in a 12-hour period and absolute neutrophil count < 0.5 x 10e9/L on the same day of the fever or the day after. | End of study

SECONDARY OUTCOMES:
Percentage of patients developing adverse events and/ or changes in laboratory values. | End of study
Incidence of neutropenia defined as absolute neutrophil count < 0.5 x 10e9/L not associated with fever | End of study
Incidence of need for IV anti-infectives and days of admission, as a result of neutropenia | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Raman Rao, MD, Study Director — Shantha Biotechnics Limited, Hyderabad, India
Locations (7):
- India (7):
  - Indo American Cancer Institute and Research Centre, Hyderabad, Andhra Pradesh
  - Nizam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Vedanta Institute of Medical Sciences, Ahmedabad, Gujarat
  - Lakeshore Hospital and Research Center, Kochi, Kerala
  - Regional Cancer Centre, Trivandrum, Kerala
  - Seth Ramdas Shah Memorial Hospital, Pune, Maharashtra
  - SMS Medical College and Hospital, Jaipur, Rajasthan